CLINICAL TRIAL: NCT02859701
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single Ascending and Multi Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AK002 in Healthy Participants
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AK002 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK002-002
Record Dates: First submitted 2016-07-13; First posted 2016-08-09 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Healthy
MeSH Terms: interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AK002 (Experimental): AK002 will be administered as an intravenous (IV) infusion in 8 cohorts of single escalating doses and two cohorts with multiple doses
  Interventions: Drug: AK002
- Placebo (Placebo Comparator): Placebo administered as anl IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AK002 — IV AK002
  Arms: AK002
Other: Placebo
  Arms: Placebo

SUMMARY:
Single-centre, randomised, double blind, placebo controlled, single ascending dose study and multiple dose study. AK002 will be administered as an intra-venous (IV) infusion in eight cohorts of single escalating doses and two cohorts with multiple doses. The study will comprise of 3 parts: Part A (Cohorts 1 - single ascending dose); Part B (Cohorts 2 to 9 - single ascending dose); Part C (Cohorts 10 and 11 - multiple dose).

DETAILED DESCRIPTION:
Participants who meet all inclusion and none of the exclusion criteria will be enrolled in the study. Safety and tolerability will be evaluated throughout the study. Blood sampling for PK and PD analysis will be also collected during the course of the study.

Up to approximately 48 participants will be enrolled in the study. Participants will be screened from -28 days prior to dose administration.

In parts A and B, participants will be admitted to the unit on Day -1 and will remain confined to the clinic until completion of Day 4 procedures. On Day 1, participants will receive a single dose of AK002 or placebo and complete study procedures. Participants will return to the clinic for follow up at Days 7, 14, 28, 56, 84 and 112 or end of study (EOS) visit.

In part C, In Part C, participants will be admitted to the unit on Day -1 and will remain confined to the clinic until completion of Day 2 procedures. On Day 1, participants will receive a dose of AK002 or placebo and complete procedures as detailed in Table 2. Participants will return to the clinic for follow up at Days 4, 7 and 14, and on Day 28 participants will receive a second dose of study drug (AK002 or a corresponding placebo) and will remain confined to the clinic until completion of the Day 29 procedures. Participants will return to the clinic for follow up at Days 31, 35, 42, 56, 84 and 112 or end of study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy volunteers, age at screening 18 to 65 years, inclusive.
2. Determined by the Investigator to be in good health, as documented by medical history, physical examination (including, but not limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, clinical laboratory assessments, and by general observations.
3. Participants must weigh at least 50 kg and have a Body Mass Index (BMI) between 18 and 30 kg/m2 Inclusive.
4. Participants must have clinical laboratory values within <1.5 x upper limit of normal (ULN) as specified by the testing laboratory, unless deemed not clinically significant by the Investigator.
5. Consumed an average of no more than 3 drinks per day within the 6 months prior to administration of study drug (beer [284 mL], wine [125 mL] or distilled spirits [25 mL]).
6. Participants must have a negative urine drug screen /alcohol breath test at screening and Day -1.
7. Stool sample negative for parasites.
8. Participants must have the ability and willingness to attend the necessary visits to the study centre.
9. Written informed consent signed prior to entry into the study.
10. Participants must be able to communicate effectively with the study site personnel.
11. Participants using highly effective, double barrier contraception (both male and female partners) during the study and for 90 days following the dose of AK002

Exclusion Criteria:

1. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
2. The participant has any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will complete the study.
3. The participant has evidence of any medical or surgical disease or condition which, in the opinion of the Investigator, might compromise the haematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, skeletal, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of AK002, or would place the participant at increased risk.
4. The participant has a history of cancer, except basal cell carcinoma which has been in remission for at least 5 years prior to Day 1
5. Use of any new drugs (including prescription and over-the-counter drugs and herbal supplements) within 1 week or 5 half-lives (whichever is longer), prior to administration of study drug.
6. Use of any prescription medication or neutraceuticals within 30 days of randomization.
7. Use of over-the counter medication (with the exception of paracetamol), vitamin supplements, or herbal medicines within 7 days of randomization.
8. Participants who initiated immunotherapy 90 days or more before the Screening visit and have been on a monthly regimen for allergy prevention or treatment may be considered for inclusion,
9. Use of immunosuppressants, oral corticosteroids, angiotensin converting enzyme (ACE) inhibitors or beta blockers within 2 weeks or 5 half-lives (whichever is longer), prior to Screening.
10. Any clinically significant laboratory abnormality or ECG.
11. The participant has a known hypersensitivity to any component of the formulation of AK002.
12. Absolute neutrophil count <1500/microliter.
13. Aspartate aminotransferase (AST) or alanine transaminase (ALT) >1.5 x ULN unless deemed not clinically significant by Investigator discretion.
14. The participant has history or presence of alcoholism or drug abuse within the 2 years prior to the first study drug administration, or is unwilling to agree to abstain from alcohol limitations and drugs throughout the study.
15. The participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 3 months prior to Check-in (Day -1). Cotinine urine test is positive at Screening or Check-in (Day -1).
16. The participant has poor peripheral venous access.
17. Blood donation or significant blood loss (more than 500 mL) within 60 days
18. Plasma donation within 7 days prior to Day 1.
19. Administration of Investigational Product (IP) in another trial within 30 days prior to the first study drug administration (or within 5 half lives of the drug, whichever is longer).
20. Females who are pregnant or lactating or intend to become pregnant before, during, or within 90 days after participating in this study; or intending to donate ova during such time period.
21. Surgery within the past three months prior to the first study drug administration determined by the PI to be clinically relevant.
22. Failure to satisfy the PI of fitness to participate for any other reason.
23. History of severe allergic or anaphylactic reactions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-08; Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AK002 as assessed by incidence, nature and severity of AEs and SAEs. | Screening to day 112

SECONDARY OUTCOMES:
Evaluate pharmacokinetic parameter AUC for AK002. | Baseline to Day 112
Change from baseline of absolute peripheral blood counts of eosinophils. | baseline to Day 112
Change from baseline of absolute peripheral blood counts of basophils. | baseline to Day 112
Changes in serum tryptase levels | baseline to Day 112
Evaluate pharmacokinetic parameter CMAX for AK002. | baseline to day 112
Changes in Eosinophilic Cationic protein levels | Baseline to day 112

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MBBS PhD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network Limited, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Undecided